CLINICAL TRIAL: NCT07023315
Title: A Randomized, Double-blind, Phase III Clinical Study Comparing the Efficacy and Safety of Cadonilimab Plus Oxaliplatin and Tegafur-Gimeracil-Oteracil Potassium (SOX) Versus Placebo Plus SOX as Perioperative Treatment for Patients With Resectable Gastric and Gastroesophageal Junction (G/GEJ) Adenocarcinoma
Brief Title: A Phase III Clinical Study of Cadonilimab Plus SOX as Perioperative Treatment for Patients With Resectable G/GEJ Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104-310
Record Dates: First submitted 2025-06-10; First posted 2025-06-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cadonilimab+SOX (Experimental): Cadonilimab plus Oxaliplatin and Tegafur-Gimeracil-Oteracil Potassium (SOX)
  Interventions: Drug: Cadonilimab; Drug: SOX chemotherapy
- Placebo+SOX (Placebo Comparator): Placebo plus Oxaliplatin and Tegafur-Gimeracil-Oteracil Potassium (SOX)
  Interventions: Drug: SOX chemotherapy; Drug: Placebo

INTERVENTIONS:
Drug: Cadonilimab — Anti-PD-1/ CTLA-4 tetrameric bispecific antibody
  Arms: cadonilimab+SOX
Drug: SOX chemotherapy — A combination treatment made up of oxaliplatin and tegafur-gimeracil-oteracil potassium
Drug: Placebo — Placebo
  Arms: Placebo+SOX

SUMMARY:
This study investigates treatment of cadonilimab or placebo combined with SOX chemotherapy (oxaliplatin + tegafur-gimeracil-oteracil potassium) given before surgery (neoadjuvant) and cadonilimab or placebo combined with SOX chemotherapy after surgery (adjuvant), will work and be safe for the treatment of resectable (removable by surgery) gastric or gastroesophageal cancer.

DETAILED DESCRIPTION:
This trial is a Phase 3 study. All patients are resectable gastric or gastroesophageal junction adenocarcinoma, Eastern Cooperative Oncology Group (ECOG) performance status 0-1.The purpose of this study is to evaluate the efficacy and safety of cadonilimab combined with chemotherapy for perioperative treatment of resectable gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed gastric or gastroesophageal junction adenocarcinoma with resectable disease (clinical stage T3-4aN+M0 or T4bNanyM0 per AJCC 8th edition).
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment.
3. Has life expectancy of at least 6 months.
4. Availability of tumor sample prior to study entry.
5. Patients must undergo radical surgery.
6. Has adequate organ function.

Exclusion Criteria:

1. Patients with unresectable locally advanced disease or distant metastasis.
2. Histopathology or cytology confirmed other pathological types, such as adenosquamous cell carcinoma, squamous cell carcinoma, or GI stromal tumor.
3. Current or prior use of immunosuppressive medication within 14 days before randomization.
4. Has received prior anti-cancer therapy for the current malignancy.
5. Has an active infection requiring systemic therapy.
6. Contra-indication to any of the study drugs.
7. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years.
8. Has an active autoimmune disease that has required systemic treatment in past 2 years.
9. Known active Hepatitis B or Hepatitis C virus infection.
10. Has had an allogenic tissue/solid organ transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 5 years
  EFS is the time from date of randomization until the date of disease progression or death.
Pathological Complete Response (pathCR) Rate | Up to approximately 2 years
  PathCR rate is defined as the percentage of participants having a pathCR assessed by the investigators.
  PathCR is defined as no invasive disease within an entirely submitted and evaluated gross lesion, and histologically negative nodes.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 10 years
  Overall survival is length of time from randomization until the date of death due to any cause.
Disease-free Survival (DFS) | Up to 5 years
  DFS is defined as the time from post-surgery baseline scan until the first occurrence of local or distant recurrence or death from any cause.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to 5 years
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Provincial Tumor Hospital, Tianjin, Tianjin Municipality